CLINICAL TRIAL: NCT00686062
Title: Adaptation and Implementation of a Prenatal Genetic Testing Decision-Assisting Tool for Clinical Use
Brief Title: Evaluation of a Decision Assisting Tool for Prenatal Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Miriam Kuppermann, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H8937-16337; AHRQ Grant # R18-HS10214
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Pregnancy
Keywords: Prenatal testing; Amniocentesis; Decision making; Down syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Women in this arm view the interactive, computerized, prenatal testing decision tool (PT Tool) we created.
  Interventions: Other: PT Tool - interactive, computerized, prenatal testing decision tool
- 2 (Active Comparator): Women in this arm view the age-appropriate computerized version of the educational pamphlet on prenatal testing developed and distributed by the State of California
  Interventions: Other: Control - computerized age-appropriate prenatal testing educational brochure

INTERVENTIONS:
Other: Control - computerized age-appropriate prenatal testing educational brochure — Computerized version of the age-appropriate prenatal testing educational brochure distributed by the State of California.
  Arms: 2
Other: PT Tool - interactive, computerized, prenatal testing decision tool — An interactive, computerized prenatal testing decision-assisting tool (PT Tool).
  Arms: 1

SUMMARY:
This is a randomized study of an interactive, computerized descision-assisting tool for prenatal testing decision making (PT Tool) versus standard educational booklets distributed to all pregnant women by the State of California (control). We hypothesize that, compared to controls, women randomized to view PT Tool will have greater knowledge about prenatal testing and its potential outcomes and better risk comprehension, and that they will be more satisfied with the intervention and have lower decisional conflict.

DETAILED DESCRIPTION:
We will evaluate the tool in a randomized controlled trial among 500 patients receiving prenatal care at one of the obstetrics clinics and practices affiliated with the University of California at San Francisco (UCSF), San Francisco General Hospital (SFGH), Kaiser San Francisco, or California Pacific Medical Center (CPMC). After completing a baseline questionnaire, participants will be randomized to view either a control or intervention group. Patients assigned to the control group will view the computerized version of the age-appropriate educational pamphlet concerning prenatal testing developed by the State of California. Patients assigned to the intervention group will use the computerized decision support tool/educational module which provides important background information about chromosomal abnormalities, and patient-tailored information about the advantages and limitations of diagnostic testing.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at less than 24 gestational weeks

Exclusion Criteria:

* Not able to speak English or Spanish

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 494
Dates: Start 2001-04; Primary Completion 2003-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kuppermann, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Kuppermann M, Norton ME, Gates E, Gregorich SE, Learman LA, Nakagawa S, Feldstein VA, Lewis J, Washington AE, Nease RF Jr. Computerized prenatal genetic testing decision-assisting tool: a randomized controlled trial. Obstet Gynecol. 2009 Jan;113(1):53-63. doi: 10.1097/AOG.0b013e31818e7ec4. PMID 19104360